CLINICAL TRIAL: NCT00806754
Title: Investigation of the Efficacy and Safety of Concomitant Administration of Ciclesonide Nasal Spray and Azelastine Nasal Spray in Patients (18 Years or Older) With Perennial Allergic Rhinitis (PAR) Not Adequately Controlled on an Intranasal Corticosteroid or Antihistamine Monotherapy
Brief Title: Investigation of the Efficacy and Safety of Concomitant Administration of Ciclesonide Nasal Spray and Azelastine Nasal Spray in Patients (18 Years or Older) With Perennial Allergic Rhinitis (PAR) Not Adequately Controlled on an Intranasal Corticosteroid or Antihistamine Monotherapy (BY9010/M1-490)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/M1-490
Record Dates: First submitted 2008-12-10; First posted 2008-12-11 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Perennial Allergic Rhinitis; Ciclesonide; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — azelastine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Ciclesonide nasal spray (50 mcg/spray, one spray per nostril) and placebo azelastine nasal spray ( two sprays per nostril) administered twice daily approximately 1 minute apart, once in the morning and 12 hours later, in the evening.
  Interventions: Drug: Ciclesonide nasal spray + placebo Azelastine
- 2 (Active Comparator): Ciclesonide nasal spray (50 mcg/spray, one spray per nostril) and azelastine nasal spray (137 mcg/spray, two sprays per nostril) administered twice daily approximately 1 minute apart, once in the morning and 12 hours later, in the evening.
  Interventions: Drug: Ciclesonide nasal spray + Azelastine

INTERVENTIONS:
Drug: Ciclesonide nasal spray + placebo Azelastine — Ciclesonide nasal spray 50 mcg + Placebo Azelastine
  Arms: 1
Drug: Ciclesonide nasal spray + Azelastine — Ciclesonide nasal spray 50 mcg + Azelastine 137 mcg
  Arms: 2

SUMMARY:
* The primary objective of this study is to evaluate the efficacy of the concomitant administration of ciclesonide nasal spray and azelastine nasal spray versus ciclesonide nasal spray alone in patients (18 years or older) with perennial allergic rhinitis (PAR) not adequately controlled on an intranasal corticosteroid or antihistamine monotherapy
* The secondary objective is to investigate the safety of the concomitant administration of ciclesonide nasal spray and azelastine nasal spray

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older at the B0 Visit.
2. General good health, and free of any concomitant conditions or treatment that in the investigator's judgment could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the trial.
3. A history of PAR for a minimum of two years immediately preceding the Screening Visit (B0). The PAR must have been of sufficient severity to require treatment(continuous or intermittent) in the past with intranasal corticosteroids and/or antihistamines and, in the investigator's judgment, experienced less than complete symptom alleviation on this prior therapy. In addition, the patient is again expected to require treatment throughout the study period.
4. A demonstrated sensitivity to at least one allergen known to induce PAR through a standard prick test within one year of study start. A positive test is defined as a wheal diameter at least 3 mm larger than the control (saline) wheal for the prick test. Documentation of a positive result within 12 months prior to the Screening Visit (B0) is acceptable.
5. Females of childbearing potential currently using contraception must continue to use a medically reliable method of contraception for the entire study duration(e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection).Females who are not sexually active must agree to use double-barrier protection should they become active during the course of the study. Women of childbearing potential, or less than 1 year postmenopausal, will require a negative plasma pregnancy test at the Screening Visit (B0). Females will be considered to be of non-child-bearing potential and will not require a urine pregnancy test if at least one of the following apply:

   * More than one year post-menopausal
   * Had a hysterectomy
   * Had bilateral ovariectomy or salpingectomy or tubal ligation
   * Has congenital sterility
6. Patients on intranasal corticosteroids and antihistamines should be on a stable dose for at least 4 weeks.
7. Patients must complete a 24-hour reflective total nasal symptom assessment at the Screening Visit (B0) and score a total of 6 or greater (out of 12).

Exclusion Criteria:

1. Pregnancy, nursing, or plans to become pregnant or donate gametes (ova or sperm) for in vitro fertilization during the study period or for 30 days following the study period.
2. History of physical findings of nasal pathology, including nasal polyps (within the last 60 days) or other clinically significant respiratory tract malformations, recent nasal biopsy (within the last 60 days), nasal trauma, or surgery and atrophic rhinitis or rhinitis medicamentosa (within the last 60 days).
3. Participation in any investigational drug trial within the 30 days preceding the Screening Visit.
4. A known hypersensitivity to any intranasal corticosteroid, antihistamine or any of the excipients in the formulation.
5. History of a respiratory infection or disorder [including, but not limited to bronchitis, pneumonia, the common cold, acute or chronic sinusitis, flu, severe acute respiratory syndrome (SARS)] within the 14 days preceding the Screening Visit, or development of a respiratory infection during the Screening Period.
6. History of alcohol or drug abuse within the preceding two years.
7. History of a positive test for HIV, hepatitis B or hepatitis C.
8. Active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of b-agonists; intermittent use of b-agonists is acceptable.
9. Use of any prohibited concomitant medications within the prescribed (per protocol) time since last dose period prior to the Screening Visit (B0) and during entire treatment duration.
10. Use of antibiotic therapy for acute conditions within 14 days prior to the Screening Visit (B0). Low doses of antibiotics taken for prophylaxis are permitted if the therapy was started prior to the Screening Visit AND is expected to continue throughout the trial.
11. Initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the Screening Visit AND use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
12. Non-vaccinated exposure to or active infection with, chickenpox or measles within the 21 days preceding the Screening Visit (B0).
13. Exposure to systemic corticosteroids for any indication, chronic or intermittent (e.g.: contact dermatitis), during the past 2 months, or presence of an underlying condition that can reasonably be expected to require treatment with corticosteroids during the course of the study.
14. Use of topical corticosteroids in concentrations in excess of 1% hydrocortisone for dermatological conditions during the past 1 month, or presence of an underlying condition that can reasonably be expected to require treatment with such preparations during the course of the study.
15. History of epilepsy or seizures (excluding febrile seizures).
16. History of coronary artery disease, uncontrolled hypertension, or other clinically significant cardiovascular disease.
17. Patients using combination treatment for allergic rhinitis (e.g. intranasal corticosteroid and antihistamine).
18. Have any of the following conditions that are judged by the investigator to be clinically significant and/or affect the subject's ability to participate in the clinical trial, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult:

    * Impaired hepatic function including alcohol-related liver disease or cirrhosis;
    * History of ocular disturbances e.g. glaucoma or posterior subcapsular cataracts;
    * Any systemic infection;
    * Hematological, hepatic, renal, endocrine (except for controlled diabetes mellitus or postmenopausal symptoms or hypothyroidism);· Gastrointestinal disease;
    * Malignancy (excluding basal cell carcinoma).
19. Clinical site employees and their immediate relatives are excluded from study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Average of AM and PM patient-reported reflective Total Nasal Symptom Score (TNSS) over the four weeks of treatment | 4 weeks

SECONDARY OUTCOMES:
Total physician-assessed nasal symptoms score (PNSS) at Endpoint | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (35):
- United States (35):
  - Altana/Nycomed, Encinitas, California
  - Altana/Nycomed, Los Angeles, California
  - Altana/Nycomed, Mission Viejo, California
  - Altana/Nycomed, San Diego, California
  - Altana/Nycomed, San Jose, California
  - Altana/Nycomed, Colorado Springs, Colorado
  - Altana/Nycomed, Denver, Colorado
  - Altana/Nycomed, Lakewood, Colorado
  - Altana/Nycomed, Gainesville, Georgia
  - Altana/Nycomed, Savannah, Georgia
  - Altana/Nycomed, Stockbridge, Georgia
  - Altana/Nycomed, Overland Park, Kansas
  - Altana/Nycomed, Metairie, Louisiana
  - Altana/Nycomed, Shreveport, Louisiana
  - Altana/Nycomed, Bethesda, Maryland
  - Altana/Nycomed, North Dartmouth, Massachusetts
  - Altana/Nycomed, Novi, Michigan
  - Altana/Nycomed, Rolla, Missouri
  - Altana/Nycomed, Papillion, Nebraska
  - Altana/Nycomed, Skillman, New Jersey
  - Altana/Nycomed, Raleigh, North Carolina
  - Altana/Nycomed, Cincinnati, Ohio
  - Altana/Nycomed, Sylvania, Ohio
  - Altana/Nycomed, Ashland, Oregon
  - Altana/Nycomed, Medford, Oregon
  - Altana/Nycomed, Portland, Oregon
  - Altana/Nycomed, Pittsburgh, Pennsylvania
  - Altana/Nycomed, Upland, Pennsylvania
  - Altana/Nycomed, Charleston, South Carolina
  - Altana/Nycomed, Dallas, Texas
  - Altana/Nycomed, San Antonio, Texas
  - Altana/Nycomed, South Burlington, Vermont
  - Altana/Nycomed, Newport News, Virginia
  - Altana/Nycomed, Richmond, Virginia
  - Altana/Nycomed, Milwaukee, Wisconsin

REFERENCES:
- See also: BY9010_M1-490 Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4544&filename=BY9010_M1-490%20Synopsis.AZCT.com%20posting.pdf